CLINICAL TRIAL: NCT00083577
Title: UARK 98-003, A Phase II Pilot Study of Anti-Angiogenesis Therapy Using Thalidomide in Patients With Multiple Myeloma
Brief Title: Anti-Angiogenesis Therapy Using Thalidomide in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UARK 98-003
Record Dates: First submitted 2004-05-25; First posted 2004-05-27 (Estimated); Last update posted 2010-07-02 (Estimated); Status verified 2010-07

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Thalidomide; Anti-Angiogenesis
MeSH Terms: conditions — Multiple Myeloma | interventions — Thalidomide

INTERVENTIONS:
Drug: Thalidomide

SUMMARY:
The purpose of this research is to study how helpful thalidomide is in controlling the myeloma disease and to study any side effect resulting from thalidomide.

DETAILED DESCRIPTION:
Patients will receive thalidomide in the oral form (by mouth). Then the dose of thalidomide will be increased each week until week 7 as long as there are no significant side effects. After week 7, patients will continue to receive thalidomide as long as there is no toxicity requiring the treatment to be stopped and as long as there is no evidence of rapid tumor growth during the treatment with thalidomide.

Routine physical examinations and blood tests will be done to monitor the effect of treatment and the toxicities encountered, if any, and provide the available treatments for side effects accordingly. Blood tests will be done once a month for the first six months of receiving thalidomide.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a confirmed diagnosis of previously treated, active multiple myeloma
* Myeloma protein should be evident from which to evaluate response
* Must be 18 years of age or older. Women of childbearing age and fertile men must use a medically acceptable means of birth control while on study and for 6 months thereafter.
* Patients must sign an informed consent to participate in this study, and be fully aware of the known teratogenic potential of this drug
* Patients must have a total white blood cell count of 2,000 K/microliters. Patients may be anemic or thrombocytopenic provided this is felt to be due to extensive marrow involvement with myeloma
* Patients must have adequate liver function as demonstrated by a direct bilirubin of < or = 2.0 mg/dL.

Exclusion Criteria:

* Patients must not have an active infection requiring parenteral antibiotics
* No other concurrent therapy for myeloma is permitted while on Thalidomide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 1998-02; Study Completion 2005-05

PRIMARY OUTCOMES:
To determine tumor response, overall and progression free survival following thalidomide therapy in patients with multiple myeloma

SECONDARY OUTCOMES:
To determine toxicities associated with thalidomide in patients with multiple myeloma

CONTACTS AND LOCATIONS:
Overall Officials: Bart Barlogie, M.D., Principal Investigator — UAMS
Locations (1):
- University of Arkansas for Medical Sciences/MIRT, Little Rock, Arkansas, United States

REFERENCES:
- See also: Myeloma Institute for Research & Therapy website — http://myeloma.uams.edu